CLINICAL TRIAL: NCT06774664
Title: A Randomized, Double-blind, Placebo-controlled Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SCTC21C in Subjects With Plasma Cell-driven Autoimmune Diseases
Brief Title: A Clinical Study of SCTC21C in Participants With Plasma Cell-driven Autoimmune Diseases
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCTC21C-X201
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Phase I: Dose-finding: Group 1 (Experimental): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase I: Dose-finding: Group 2 (Experimental): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase I: Dose-finding: Group 3 (Experimental): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase I: Dose-finding: Group 4 (Experimental): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase 2: Group 1 (Experimental): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase 2: Group 2 (Experimental): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase I: Dose-finding: Group 5 (Placebo Comparator): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase I: Dose-finding: Group 6 (Placebo Comparator): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase 1: Dose-finding: Group 7 (Placebo Comparator): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C
- Phase 2: Group 3 (Placebo Comparator): Drug: SCTC21C Administered SC
  Interventions: Biological: SCTC21C

INTERVENTIONS:
Biological: SCTC21C — Drug: SCTC21C Administered SC

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of SCTC21C in subjects with plasma cell-driven autoimmune diseases

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase I/II study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of multiple doses of SCTC21C in subjects with plasma cell-driven autoimmune diseases.

In phase 1 study, participants will be assigned to receive sequentially higher doses of SCTC21C to determine the recommended dose of SCTC21C for the randomized dose optimization- stage. In phase 2 study, 2 dose levels will be used. A total of 72 participants will be randomized in a 1:1:1 ration to dose 1, dose 2 or placebo groups to better understand the exposure/efficacy/toxicity relationship.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the ICF;
2. The subject has been diagnosed with IgA nephropathy through kidney tissue biopsy;
3. The subject has been on a stable and maximally tolerated dose of ACEI or ARB (or the maximum allowable dose according to the prescribing information) for at least 12 weeks prior to the first dose. Subjects using both ACEI and ARB simultaneously will not be accepted;
4. The estimated glomerular filtration rate (eGFR) calculated using the CKD-EPI formula must be ≥30 mL/min/1.73 m²;
5. During the screening period, the subject must have 24-hour proteinuria ≥1.0 g or a urine protein-to-creatinine ratio (UPCR) ≥0.75 g/g based on 24-hour urine protein;
6. All male subjects or women of childbearing potential (with a negative blood pregnancy test within 7 days prior to the first dose of investigational drug) must agree to use reliable contraception together with their partner from the time of signing the ICF until 5 months after the last dose of the study drug;
7. Understand the study procedures and voluntarily sign the informed consent form in writing.

Exclusion Criteria:

1. IgA nephropathy secondary to other diseases;
2. Any kidney disease with special pathological or clinical types, such as nephrotic syndrome, crescentic glomerulonephritis, etc.;
3. Use of systemic corticosteroids within the 3 months prior to baseline or expected use during the study period;
4. Use of systemic immunosuppressive drugs within the 3 months prior to baseline or expected use during the study period;
5. Use of other B-cell-targeting biologics or unapproved investigational biologics within the 6 months prior to baseline;
6. Patients who have experienced any of the following cardiovascular events within 24 weeks prior to baseline: myocardial infarction, unstable angina, ventricular arrhythmias, heart failure with NYHA class II or higher, stroke, etc.;
7. A history of solid organ or hematopoietic stem cell or bone marrow transplantation, or expected to undergo a transplant procedure during the treatment period with the investigational drug；
8. Currently undergoing hemodialysis or peritoneal dialysis, or expected to require hemodialysis or peritoneal dialysis during the treatment period with the investigational drug;
9. Any symptoms or signs within 30 days prior to baseline indicating an active infection (excluding the common cold), or requiring systemic anti-infective treatment, or being at high risk for infection;
10. Positive viral serology, including HIV, HCV, and HBV, etc.; Hepatitis B patients: active hepatitis or severe liver disease;
11. Currently or within the past 5 years has had malignant tumors, except for fully treated skin basal cell carcinoma, squamous cell carcinoma, cervical carcinoma in situ, or cervical intraepithelial neoplasia;
12. Known allergy to the active ingredient or excipients of the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Treatment-emergent adverse events (TEAEs), serious adverse events (SAEs). | 36 Weeks
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  Results in death Is life-threatening Requires in patient hospitalisation or prolongation of existing hospitalisation Is a congenital anomaly or birth defect Is an infection that requires treatment parenteral antibiotics Other important medical events which based on medical or scientific judgement may jeopardise the patients, or may require medical or surgical intervention to prevent any of the above.
Phase 2: Percentage change in urine protein-to-creatinine ratio (UPCR) at Week 24 compared to baseline | 24 Weeks
  UPCR is calculated by dividing the concentration of protein in urine by the urine creatinine concentration.

SECONDARY OUTCOMES:
Phase 1: Percentage change in urine protein-to-creatinine ratio (UPCR) compared to baseline | 36 Weeks
  UPCR is calculated by dividing the concentration of protein in urine by the urine creatinine concentration.
Phase 1: Percentage change in 24-hour urinary protein excretion compared to baseline | 36 Weeks
Phase 1: Percentage change in urine albumin-to-creatinine ratio (UACR) compared to baseline | 36 Weeks
  UACR is calculated by dividing the concentration of albumin in urine by the urine creatinine concentration.
Phase 1: Percentage change in eGFR compared to baseline | 36 Weeks
  eGFR is calculated using the CKD-EPI formula.
Phase 1: Change from baseline in Immunoglobulin A (IgA), Immunoglobulin M (IgM), Immunoglobulin G (IgG), etc. | 36 Weeks
Phase 1: C-max | 24 Weeks
  Maximum observed plasma concentration
Phase 1: T1/2 | 24 Weeks
  apparent terminal half-life
Phase 1: AUC0-t | 24 Weeks
  area under the plasma concentration time curve from time 0 to the time of last observed quantifiable concentration
Phase 1: Percentage of Participants With Positive Antidrug Antibody (ADA) and Neutralizing Antibody (Nab) | 36 Weeks
  Results for ADA analysis were reported.
Phase 2: Percentage change in urine protein-to-creatinine ratio (UPCR) compared to baseline | 104 Weeks
  UPCR is calculated by dividing the concentration of protein in urine by the urine creatinine concentration.
Phase 2: Percentage change in 24-hour urinary protein excretion compared to baseline | 104 Weeks
Phase 2: Percentage change in urine albumin-to-creatinine ratio (UACR) excretion compared to baseline | 104 Weeks
  UPCR is calculated by dividing the concentration of albumin in urine by the urine creatinine concentration.
Phase 2: Percentage change in eGFR compared to baseline | 104 Weeks
  eGFR is calculated using the CKD-EPI formula.
Phase 2: Change from baseline in Immunoglobulin A (IgA), Immunoglobulin M (IgM), Immunoglobulin G (IgG), etc. | 104 Weeks
Phase 2: C-max | 32 Weeks
  Maximum observed plasma concentration
Phase 2: T1/2 | 32 Weeks
  apparent terminal half-life
Phase 2: AUC0-t | 32 Weeks
  area under the plasma concentration time curve from time 0 to the time of last observed quantifiable concentration
Phase 2: Percentage of Participants With Positive Antidrug Antibody (ADA) and Neutralizing Antibody (Nab) | 104 Weeks
  Results for ADA analysis were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Principal Investigator — Peking University First Hospital, Department of Nephrology
Locations (20):
- China (20):
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Sichuan Academy of Medical Sciences - Sichuan Provincial People's Hospital, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Shandong Provincial Hospital, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning
  - Ningbo NO.2 Hospital, Ningbo
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Wuxi People's Hospital, Wuxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai
  - Yantai Yuhuangding Hospital, Yantai
  - General Hospital of Ningxia Medical University, Yinchuan